CLINICAL TRIAL: NCT03570879
Title: Analysis of Surgical Outcomes in Women Undergoing Laparoscopic Myomectomy With Morcellation or Transvaginal Extraction of Surgical Specimens
Brief Title: Laparoscopic Myomectomy With Morcellation or Transvaginal Extraction of Surgical Specimens.
Acronym: MYMOTE-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: MYMOTE-1
Record Dates: First submitted 2018-05-30; First posted 2018-06-27 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Myoma;Uterus
Keywords: Laparoscopy; Power morcellation; Transvaginal extraction
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Power morcellation: Women that underwent laparoscopic myomectomy with subsequent power morcellation of the surgical specimens.
  Interventions: Device: Power morcellation
- Transvaginal extraction: Women that underwent laparoscopic myomectomy with subsequent transvaginal extraction of the surgical specimens.
  Interventions: Procedure: Transvaginal extraction

INTERVENTIONS:
Device: Power morcellation — Power morcellation of surgical specimens after laparoscopic myomectomy.
  Groups: Power morcellation
Procedure: Transvaginal extraction — Transvaginal extraction of surgical specimens after laparoscopic myomectomy.
  Groups: Transvaginal extraction

SUMMARY:
Laparoscopic myomectomy represents the fertility-sparing gold standard approach for the management of subserosal and intramural uterine myomas: this technique allows faster recovery, less complications and improved surgical outcomes than laparotomy.

Despite these validated cornerstones of minimally invasive gynecology, the best approach for specimen retrieval is still debated. Among these approaches, surgical specimen retrieval after laparoscopic myomectomy could be performed by mini-laparotomy, by power morcellation using morcellator inserted through one of the ancillary trocars, or by transvaginal extraction through an endobag inserted at level of the posterior vaginal fornix (between the utero-sacral ligaments).

Unfortunately, mini-laparotomy has poor esthetic outcome and does not conform the current standards of minimally invasive surgery.

In addition, on 24 November 24 2014 the Food and Drug Administration updated a Safety Communication about Power Morcellation, warning against the use of laparoscopic power morcellators in the majority of women undergoing myomectomy or hysterectomy for treatment of fibroids, due to the risk of spreading an unsuspected uterine sarcoma within the abdomen and pelvis.

Considering this scenario, transvaginal extraction may represents a feasible approach for specimen retrieval. In this view, the current study aims to retrospectively compare surgical outcomes in women that underwent laparoscopic myomectomy with subsequent power morcellation (before the issuing of the abovementioned Safety Communication by the Food and Drug Administration) or transvaginal extraction (after the issuing of the abovementioned Safety Communication by the Food and Drug Administration) of the surgical specimens.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by single or multiple uterine myomas.
* Signed informed consent.

Exclusion Criteria:

* Human papilloma virus-related pathologies at pap-smear within the 12 months preceding surgery.
* Women with obliteration of the cul-de-sac.
* Women with the suspected cancer of gynecological origin.
* Women who had never experienced complete sexual intercourse before the operation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women that underwent laparoscopic myomectomy with subsequent power morcellation (before the issuing of the abovementioned Safety Communication by the Food and Drug Administration) or transvaginal extraction (after the issuing of the abovementioned Safety Communication by the Food and Drug Administration) of the surgical specimens.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Complication rate | Within 12 months after surgery.
  Number of surgical complications (Clavien-Dindo Classification)

SECONDARY OUTCOMES:
Operative time | Through study completion, an average of 10 years (retrospective analysis)
  Duration of the surgery, expressed in minutes.
Blood loss | Through study completion, an average of 10 years (retrospective analysis)
  Blood loss during the surgery, expressed in milliliters (ml).
Hospital stay | Through study completion, an average of 10 years (retrospective analysis)
  Duration of the hospitalization, expressed in days
Sexual function | 6 and 12 months after surgery.
  Sexual function evaluated by Female Sexual Function Index questionnaire, investigating quantity and quality of sex [scale total score minimum: 2 (worse outcome), maximum: 36 (best outcome)]

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Jvan Casarin, M.D., Principal Investigator — Università degli Studi dell'Insubria; Antonella Cromi, M.D., Ph.D., Study Chair — Università degli Studi dell'Insubria; Fabio Ghezzi, M.D., Study Director — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided